CLINICAL TRIAL: NCT00302913
Title: Efficacy of Adjusted Clopidogrel Dose in Patients With Insufficient Platelet Inhibition After Elective Coronary Stenting
Brief Title: Efficacy of Adjusted Clopidogrel Dose in Patients With Insufficient Platelet Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZ-BK-2005-2
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-02

CONDITIONS: Coronary Artery Disease; Drug Resistance
Keywords: Clopidogrel; Coronary Artery Disease; Dose-Response Relationship, Drug; Drug Resistance; PCI
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Drug: Adjustment of clopidogrel dose

SUMMARY:
This study is a prospective, single-center evaluation of the efficacy of clopidogrel dose adjustment in patients with insufficient platelet inhibition after elective coronary stent implantation.

DETAILED DESCRIPTION:
Background: The EXCELSIOR trial demonstrated a 7-fold increased risk for death, myocardial infarction and target vessel reintervention within 30 days in patients with platelet inhibition below median of study cohort after a bolus dose of 600 mg of clopidogrel. The median of platelet inhibition in this cohort was 14 % optical aggregation after stimulation with 5 µM ADP.

Aim: To evaluate the efficacy of clopidogrel dose adjustment in patients with insufficient platelet inhibition after elective coronary stent implantation

Methods: This prospective, single-center study will evaluate antiplatelet effects in 120 patients receiving a bolus dose of 600 mg of clopidogrel before undergoing elective coronary stent implantation. Platelet inhibition will be evaluated 24 hours, 14 and 28 days after coronary intervention using optical aggregometry (5 µM ADP) and determination of surface protein expression by flow cytometry (P-Selectin, gp55, activated GP IIb/IIIa). If 24 hours after coronary stent implantation optical aggregation is >14 %, patients will receive an additional bolus dose of 300 mg of clopidogrel, followed by a daily dose of 150 mg for at least 28 days. If optical aggregation at this point of time is ≤14 % patients will receive a daily dose of 75 mg of clopidogrel. No further dose adjustments during follow up will be performed.

Hypothesis: Adjustment of clopidogrel dose in patients with insufficient platelet inhibition determined by optical aggregometry will provide a comparable antiplatelet effect as in patients with sufficient platelet inhibition after coronary stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary stenting
* Pretreatment with a bolus dose of 600mg of clopidogrel at least 2 hours prior to coronary stent implantation
* Pretreatment with aspirin ≥ 100 mg per day for at least 7 days
* Age > 18 years
* Written consent

Exclusion Criteria:

* Troponin T on admission > 0.03 ng/mL
* Myocardial infarction or fibrinolytic therapy within the previous 14 days
* Cardiogenic shock
* Contraindication for aspirin or clopidogrel
* Oral anticoagulation
* Pretreatment with heparin or a thienopyridine within the previous 14 days
* Use of a GP IIb/IIIa-receptor antagonist during PCI
* Platelet count < 100.000/µl
* Severe disorders of the coagulation system
* Severe impairment of liver or kidney function
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-12; Study Completion 2006-06

PRIMARY OUTCOMES:
Antiplatelet effect after fourteen and twenty-eight days determined by optical aggregometry after stimulation with ADP

SECONDARY OUTCOMES:
Antiplatelet effect after fourteen and twenty-eight days determined by flow cytometric evaluation of surface protein expression after stimulation with ADP
Major cardiac events within thirty days (death, myocardial infarction, target vessel reintervention)
Bleeding and vascular access site complications within thirty days
Drug-drug interaction of clopidogrel with concomitant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Josef Neumann, MD, Study Director — Heart Center Bad Krozingen, Germany
Locations (1):
- Heart Center Bad Krozingen,, Bad Krozingen, Germany